CLINICAL TRIAL: NCT03189966
Title: Effect of Different Truncal Blocks Under Ultrasound-Guidance on Pain Management After Open Reduction of Pediatric Developmental Dysplasia of the Hip: a Randomized Trial
Brief Title: Truncal Blocks for Pediatric With Developmental Dysplasia of the Hip Undergoing Open Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, congcong huang, Department of Anesthesiology, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18
Record Dates: First submitted 2017-04-26; First posted 2017-06-16 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Developmental Dysplasia of the Hip (DDH)
Keywords: transversalis fascia plane block; quadratus lumborum block; ultrasound-guided; Developmental Dysplasia of the Hip; postoperative analgesia
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group T (Experimental): Patients in transversalis fascia plane block group(Group T) will receive ultrasound-guided transversalis fascia plane block using0.3% ropivacaine(0.8 ml/kg) after general anesthesia
  Interventions: Procedure: transversalis fascia plane block
- Group Q (Experimental): Patients in quadratus lumborum block group（Group Q） will receive ultrasound-guided quadratus lumborum block using0.3%ropivacaine(0.8 ml/kg).after general anesthesia.
  Interventions: Procedure: quadratus lumborum block
- Group C (No Intervention): Patients in the third group as control (Group C)receive no nerve block.Patients will be extubated based on clinical criteria.

INTERVENTIONS:
Procedure: transversalis fascia plane block — With the patient in a supine position, the needle is advanced from the anterior using an in-plane technique. A linear ultrasound probe is orientated transversely over the lateral abdomen between the iliac crest and the costal margin. Local anesthetic is injected to separate the transversalis fascia from the transversus muscle. The correct needle position was confirmed by injection of 2 ml of normal saline solution that was spreading anterio-posteriorly between the anterior border of QLM and its fascia, in addition to a minimal anterior spread in TAP plane. After negative aspiration, 0.8 ml/Kg of ropivacaine 0.3%was injected.
  Arms: Group T
Procedure: quadratus lumborum block — The needle is directed in the posterior to anterior orientation with the practitioner standing behind the patient. The triangular quadratus lumborum (QL) muscle is adherent to the apex of the transverse process of L3 vertebra. Using the Shamrock method, the needle penetrates the QL muscle with an in-plane approach from the posterior side of the ultrasound probe. The target point is the inter fascial plane between the QL and the psoas major muscle just deep to the transversalis fascia, in order to lessen the risk of unintentional penetration of the peritoneal cavity contrary to the technique. The correct needle position was confirmed by injection of 2 ml of normal saline solution that was spreading anterio-posteriorly between the QL and the psoas major muscle. After negative aspiration, 0.8 ml/Kg of ropivacaine 0.3%was injected.
  Arms: Group Q

SUMMARY:
The aim of the study is to evaluate the effectiveness of ultrasound-guided transversalis fascia plane block (TFPB) and quadratus lumborum block (QLB) on post-operative analgesia in pediatric patients with Developmental Dysplasia of the Hip (DDH)under going open reduction surgeries（Salter acetabular osteotomy，combined with proximal femoral rotation osteotomy）.The effectiveness of TFPB/QLB for perioperative analgesia in lumbar nerves (L1) innervated surgery have been demonstrated in recent studies. However, this regional technique rarely applied to children.The objective of our research is to assess the quality of postoperative analgesia in pediatric patients who had received a preoperative TFPB/QLB for hip surgery.

DETAILED DESCRIPTION:
90 pediatric patients(age 2-10years) in the BeiJing Ji Shui Tan Hospital and The Second Affiliated Hospital of Wen Zhou Medical University with American Society of Anesthesiologists (ASA) physical status I or II, who are scheduled to undergo open reduction surgeries （Salter acetabular osteotomy，combined with proximal femoral rotation osteotomy）are selected and divided into 3 equal groups with 30 subjects.The consent forms are approved by the institutional Ethics Committee.

Inclusion Criteria: Pediatric patients between 2 years to 10 years with DDH, scheduled for unilateral open reduction surgeries（Salter acetabular osteotomy，combined with proximal femoral rotation osteotomy）.

Exclusion Criteria:Patients will be excluded if participants meet any of the following criteria:patients with known allergy to local anaesthetics, mental disability, peripheral neuropathy, a coagulopathy disorder,localized infection in the area, and any reason cause reoperation.

Electrocardiogram, non-invasive blood pressure, pulse oximetry, temperature,capnography, and end tidal anesthetic concentration values are monitored in patients Parental presence will be allowed if requested for the induction of anesthesia. Pediatrics without vein access will receive general anesthesia which induces with 8% sevoflurane in 70% nitrous oxide and 30% oxygen, via a facemask. When loss of consciousness is achieved,investigators need to establish vein access routinely.Intravenous induction for general anesthesia with endotracheal intubation is commenced using intravenous propofol 3 mg/kg, cis-atracurium 0.2 mg/kg,fentanyl 2. ug/kg. Anesthesia will be maintained using remifentanyl, and a volatile anesthetic(sevoflurane). The inhaled concentration of sevoflurane will be adjusted to maintain hemodynamic stability, which is defined as a change in systolic blood pressure and heart rate of no more than 20% of baseline parameters. The use of opioids during the perioperative periods at the discretion of the anesthetist. Some anesthetists administer opioids preemptively, however, in the majority of cases the decision is based on the cardiovascular response to stimulation; an increase in heart rate of 10% from baseline is usually interpreted as insufficient analgesia and is treated with opioids. Patients will be given either fentanyl in doses of 1-2mcg/kg, remifentanil as continuous infusion 0.01-0.03 mcg/ (kg.min) or a combination of these.

TFPB group Patients in transversalis fascia plane block group(Group T) will receive ultrasound-guided transversalis fascia plane block using0.3% ropivacaine(0.8 ml/kg) after general anesthesia. A high-frequency probe (Sono-Site HFL50x, 15- 6 MHz, 55-mm broadband linear array) connected to an S-nerve ultrasound machine((Sonosite Inc,Bothell, WA, USA) was positioned with a transverse orientation, between iliac crest and costal margin.With the patient in a supine position, the needle is advanced from the anterior using an in-plane technique. A linear ultrasound probe is orientated transversely over the lateral abdomen between the iliac crest and the costal margin. The external oblique, internal oblique,and transversus abdominis muscles are imaged, and the more posterior transversus aponeurosis is isolated from these muscles.The reflection of the peritoneum curving away from the muscles from anterior to posterior, and the perinephric fat, which lies behind the peritoneum and deep to the transversalis fascia, are both identified. The perinephric fat is generally more prominent closer to the iliac crest. The quadratus lumborum is identified medial to the aponeurosis of the transversus abdominis. The end point is more visible if the needle is passed through the posterior''tail'' of the transversus muscle, as the transversus aponeurosis is thinner and less distinct as a separate layer. After passing through the deep surface of transversus abdominis muscle, local anesthetic is injected to separate the transversalis fascia from the transversus muscle. The correct needle position was confirmed by injection of 2 ml of normal saline solution that was spreading anterio-posteriorly between the anterior border of QLM and its fascia, in addition to a minimal anterior spread in TAP plane. After negative aspiration, 0.8 ml/Kg of ropivacaine 0.3%was injected.

QLB group Patients in quadratus lumborum block group（Group Q） will receive ultrasound-guided quadratus lumborum block using 0.3% ropivacaine(0.8 ml/kg).after general anesthesia.The TFPB is performed with the patient in the lateral position using a curvilinear low-frequency ultrasound probe.This is orientated transversely at the posterior axillary line between the iliac crest and the costal margin using a 22G 100-mm needle.The needle is directed in the posterior to anterior orientation with the practitioner standing behind the patient. The triangular quadratus lumborum (QL) muscle is adherent to the apex of the transverse process of L3 vertebra.Using the Shamrock method, a new transmuscular quadrates lumborum block technique, developed by Børglum (British Journal of Anaesthesia, 2013), the needle penetrates the QL muscle with an in-plane approach from the posterior side of the ultrasound probe. The target point is the interfascial plane between the QL and the psoas major muscle just deep to the transversalis fascia, in order to lessen the risk of unintentional penetration of the peritoneal cavity contrary to the technique. The correct needle position was confirmed by injection of 2 ml of normal saline solution that was spreading antero-posteriorly between the QL and the psoas major muscle. After negative aspiration, 0.8 ml/Kg of ropivacaine 0.3%was injected.

Control group Patients in the third group as control (Group C) receive no nerve block.Patients will be extubated based on clinical criteria.

Patients will then be transported to the post-operative anesthesia care unit (PACU) after extubation.All pediatric patients will receive 6-hourly paracetamol post-operatively for two days and receive sufentanyl via nurse-controlled analgesia (NCA) or patient-controlled analgesia (PCA). The prescription of post-operative NCA/PCA is also at the discretion of the anesthetist. Children under the age of 6 years will receive sufentanyl via NCA continuously at a rate of 2 mcg/(kg.48h) with a bolus option of 0.01 mcg/kg every 15 minutes.Older children will receive sufentanyl via PCA continuously at a rate of 2 mcg/( kg.48h) with a bolus option of 0.01 mcg/kg every 15 minutes.

Data collection will include the type of procedure, age, weight, type of truncal block (QLB group vs TFPB vs control).Primary outcome was the FLACC (ie, the Face, Legs, Activity, Consolability Scale) score of patients in the PACU and at 2h, 4h, 8h, 12h, 24h, 48h postoperatively. Secondary outcomes included intraoperative MBP and HR at the endpoints of Salter acetabular osteotomy(T1), femoral rotation osteotomy (T2), and anterior superior iliac spine osteotomy (T3) during the surgery; intraoperative opioid consumption (i.e., fentanyl and remifentanil); duration of the surgery; postoperative fentanyl consumption in the PACU, postoperative morphine consumption in the ward; the length of PACU stay; the time until first press of NCA/PCA pump and the total counts number of pressing the pump; length of hospital stay; complications (e.g., immediate complications such as vessel puncture and possible undesirable effects such as hypotension, bradycardia, epidural local anesthetic spread, or postoperative nausea and vomiting). The number of doses of rescue analgesics (morphine 0.05 mg/kg) in the postoperative period (48 h) will be recorded. Rescue treatment of postoperative nausea and vomiting,will be treated with ondansetron (0.1 mg/kg) if needed.Side effects such as pruritus will also be noted.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged between 2 years and 10 years with DDH,
* scheduled for unilateral open reduction surgeries（Salter acetabular osteotomy，combined with proximal femoral rotation osteotomy）

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

* patients with known allergy to local anaesthetics,
* mental disability,
* peripheral neuropathy,
* a coagulopathy disorder,
* localized infection in the area,
* any reason cause reoperation.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change of FLACC pain scores at different time points (at rest and at movement) | for the first 48 post-operative hours（at PACU, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 48 hours after surgery）,the analgesic effects of patients at different times need to be evaluated, both at rest and at movement
  using age-appropriate and validated tools (ie, the Face, Legs, Activity, Consolability Scale [FLACC] which evaluates the intensity of pain, ranged from 0-10, 0 means no pain and 10 means severe pain) to evaluate the change of pain scores at different time points which indirectly reflect the analgesia effect, both at rest and at movement.

SECONDARY OUTCOMES:
The analgesia effects | for the first 48 post-operative hours
  The first time (hours after surgery) and the total numbers to press the analgesia pump (numbers) will be recorded.
the rescue analgesics | for the first 48 post-operative hours
  The number of doses of rescue analgesics (morphine 0.05 mg/kg) will be recorded.
complications | for the first 48 post-operative hours
  Postoperative nausea and vomiting (the numbers of participants with nausea and vomiting), hematoma (the number of participants with hematoma), nerve injury (the number of participants with nerve injury) will be recorded
Intra-operative opioid consumptions | during the surgery, average 3 hours
  intraoperative opioid consumption ((both fentanyl and remifentanil were converted into fentanyl equivalents).
PACU fentanyl consumptions | the time of staying in postanesthesia care unit(PACU), about 30 minutes to 60 minutes after surgery
  If a pain score was >3, the patient in the PACU would receive fentanyl (iv,1 μg·kg-1), while in the surgical ward morphine (iv,0.05 mg·kg-1) was administered.
PACU fentanyl rate | the time of staying in post-anesthesia care unit(PACU), about 30 minutes to 60 minutes after surgery
  the number of patients who received the fentanyl in each group during the PACU
PACU stay | the time of staying in post-anesthesia care unit(PACU), about 30 minutes to 60 minutes after surgery
  staying period in the PACU
Hospital stay | the time of staying in hospital, average 12 days
  staying period in the hospital
Parental satisfaction score (0-10) | at 48 post-operative hours, when removed the NCA/PCA pump
  Satisfaction from all patients' guardians were surveyed with regard to the postoperative analgesia of their children at the time of the NCA/PCA pump removal

CONTACTS AND LOCATIONS:
Overall Officials: CongCong Huang, Master, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (2):
- China (2):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Second Affiliated Hospital of WenZhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ueshima H, Yoshiyama S, Otake H. RETRACTED: The ultrasound-guided continuous transmuscular quadratus lumborum block is an effective analgesia for total hip arthroplasty. J Clin Anesth. 2016 Jun;31:35. doi: 10.1016/j.jclinane.2015.12.033. Epub 2016 Mar 22. PMID 27185672 (Retraction: PMID 35393191 J Clin Anesth. 2022 Aug;79:110702; PMID 35397960 J Clin Anesth. 2022 Aug;79:110704)
- [Background] Parras T, Blanco R. Randomised trial comparing the transversus abdominis plane block posterior approach or quadratus lumborum block type I with femoral block for postoperative analgesia in femoral neck fracture, both ultrasound-guided. Rev Esp Anestesiol Reanim. 2016 Mar;63(3):141-8. doi: 10.1016/j.redar.2015.06.012. Epub 2015 Aug 22. English, Spanish. PMID 26302669
- [Background] Chin KJ, Chan V, Hebbard P, Tan JS, Harris M, Factor D. Ultrasound-guided transversalis fascia plane block provides analgesia for anterior iliac crest bone graft harvesting. Can J Anaesth. 2012 Jan;59(1):122-3. doi: 10.1007/s12630-011-9610-7. Epub 2011 Oct 19. No abstract available. PMID 22009659
- [Background] Lee S, Goetz T, Gharapetian A. Unanticipated Motor Weakness with Ultrasound-Guided Transversalis Fascia Plane Block. A A Case Rep. 2015 Oct 1;5(7):124-5. doi: 10.1213/XAA.0000000000000237. PMID 26402025
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Abdallah FW, Chan VW, Brull R. Transversus abdominis plane block: a systematic review. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):193-209. doi: 10.1097/AAP.0b013e3182429531. PMID 22286518
- [Background] Sakamoto H, Akita K, Sato T. An anatomical analysis of the relationships between the intercostal nerves and the thoracic and abdominal muscles in man. I. Ramification of the intercostal nerves. Acta Anat (Basel). 1996;156(2):132-42. doi: 10.1159/000147838. PMID 8993633
- [Background] JAMIESON RW, SWIGART LL, ANSON BJ. Points of parietal perforation of the ilioinguinal and iliohypogastric nerves in relation to optimal sites for local anaesthesia. Q Bull Northwest Univ Med Sch. 1952;26(1):22-6. No abstract available. PMID 14912259
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Hansen CK, Dam M, Bendtsen TF, Borglum J. Ultrasound-Guided Quadratus Lumborum Blocks: Definition of the Clinical Relevant Endpoint of Injection and the Safest Approach. A A Case Rep. 2016 Jan 15;6(2):39. doi: 10.1213/XAA.0000000000000270. No abstract available. PMID 26771297
- [Background] Dam M, Hansen CK, Borglum J, Chan V, Bendtsen TF. A transverse oblique approach to the transmuscular Quadratus Lumborum block. Anaesthesia. 2016 May;71(5):603-4. doi: 10.1111/anae.13453. No abstract available. PMID 27072772
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] Elsharkawy H. Quadratus lumborum block with paramedian sagittal oblique (subcostal) approach. Anaesthesia. 2016 Feb;71(2):241-2. doi: 10.1111/anae.13371. No abstract available. PMID 26750418
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838
- [Background] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Barrington MJ, Ivanusic JJ, Rozen WM, Hebbard P. Spread of injectate after ultrasound-guided subcostal transversus abdominis plane block: a cadaveric study. Anaesthesia. 2009 Jul;64(7):745-50. doi: 10.1111/j.1365-2044.2009.05933.x. PMID 19624629
- [Background] Hebbard PD. Transversalis fascia plane block, a novel ultrasound-guided abdominal wall nerve block. Can J Anaesth. 2009 Aug;56(8):618-20. doi: 10.1007/s12630-009-9110-1. Epub 2009 Jun 4. No abstract available. PMID 19495909
- [Background] Rosario DJ, Jacob S, Luntley J, Skinner PP, Raftery AT. Mechanism of femoral nerve palsy complicating percutaneous ilioinguinal field block. Br J Anaesth. 1997 Mar;78(3):314-6. doi: 10.1093/bja/78.3.314. PMID 9135313
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Lancaster P, Chadwick M. Liver trauma secondary to ultrasound-guided transversus abdominis plane block. Br J Anaesth. 2010 Apr;104(4):509-10. doi: 10.1093/bja/aeq046. No abstract available. PMID 20228188
- [Background] Weikel AM, Habal MB. Meralgia paresthetica: a complication of iliac bone procurement. Plast Reconstr Surg. 1977 Oct;60(4):572-4. PMID 909967
- [Background] Fernyhough JC, Schimandle JJ, Weigel MC, Edwards CC, Levine AM. Chronic donor site pain complicating bone graft harvesting from the posterior iliac crest for spinal fusion. Spine (Phila Pa 1976). 1992 Dec;17(12):1474-80. doi: 10.1097/00007632-199212000-00006. PMID 1471005
- [Background] Smith SE, DeLee JC, Ramamurthy S. Ilioinguinal neuralgia following iliac bone-grafting. Report of two cases and review of the literature. J Bone Joint Surg Am. 1984 Oct;66(8):1306-8. No abstract available. PMID 6386820
- [Background] Lopez-Gonzalez JM, Lopez-Alvarez S, Jimenez Gomez BM, Arean Gonzalez I, Illodo Miramontes G, Padin Barreiro L. Ultrasound-guided transversalis fascia plane block versus anterior transversus abdominis plane block in outpatient inguinal hernia repair. Rev Esp Anestesiol Reanim. 2016 Nov;63(9):498-504. doi: 10.1016/j.redar.2016.02.005. Epub 2016 Apr 8. English, Spanish. PMID 27067036
- [Derived] Huang C, Zhang X, Dong C, Lian C, Li J, Yu L. Postoperative analgesic effects of the quadratus lumborum block III and transversalis fascia plane block in paediatric patients with developmental dysplasia of the hip undergoing open reduction surgeries: a double-blinded randomised controlled trial. BMJ Open. 2021 Feb 4;11(2):e038992. doi: 10.1136/bmjopen-2020-038992. PMID 33542037

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03189966/Prot_SAP_001.pdf